CLINICAL TRIAL: NCT00497718
Title: The Effect of Chiropractic Manipulation on Spine-related Pain and Balance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Chiropractic College (Other)
Responsible Party: Dr. Cheryl Hawk, Cleveland Chiropractic College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-02142007
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Musculoskeletal Equilibrium; Back Pain
MeSH Terms: conditions — Back Pain | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Chiropractic Manipulation

SUMMARY:
The effect of chiropractic manipulation on spine-related pain and balance in older adults.

DETAILED DESCRIPTION:
Chronic pain and risk factors for falls in older adults are significant public health issues. In order to evaluate an appropriate role for chiropractic in managing these problems in the population, this pilot cohort study will take multiple measurements, both self-reported and functional, on a sample of older adults with chronic spine-related pain who are recruited from the local community and receive chiropractic care in the Cleveland Chiropractic College health center over a four-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 or older
2. spine-related pain of >3 months duration (by self-report).

Exclusion Criteria:

1. Non-ambulatory
2. chiropractic care or physical therapy within the past month (by self report)
3. contraindications to manipulation, as determined by the clinician through physical exam and x-rays (if indicated)
4. absence of indications for CMT, as determined by the clinician through history, physical exam, orthopedic tests, and static and motion palpation
5. unable to understand English adequately to complete study forms.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Test various recruitment methodologies. | Through December 2008
Describe baseline characteristics of enrolled patients. | Through December 2008
Assess patient outcomes in terms of balance, neck or back pain, and dizziness | Through December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Hawk, D.C., Ph.D., Principal Investigator — Cleveland Chiropractic College
Locations (1):
- Cleveland Chiropractic College Health Center, Kansas City, Missouri, United States